CLINICAL TRIAL: NCT04056442
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Crossover, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of Cannabidiol (CBD) as a Steroid-sparing Therapy in Steroid-dependent Crohn's Disease Patients
Brief Title: A Phase 2a Study to Evaluate the Safety, Tolerability and Efficacy of Cannabidiol as a Steroid-sparing Therapy in Steroid-dependent Crohn's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stero Biotechs Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ST-SDCD-01
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Steroid Dependent Crohn's Disease
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at a 2:1 Cannabidiol:placebo ratio. After 3 month of treatment a blinded assessor will assess the patient response.
  Cannabidiol Non-responders will be removed from the trial, and Placebo Non-responders will be switched over to Cannabidiol
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): 300 mg Cannabidiol (synthetic form) Olive Oil Solution, 5%
  Interventions: Drug: Cannabidiol , synthetic form; Drug: Placebo
- Placebo (Placebo Comparator): Olive Oil Solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol , synthetic form — Cannabidiol ( synthetic form)
  Arms: Cannabidiol
Drug: Placebo — Olive Oil Solution, 5%

SUMMARY:
Treatment will start with dose escalation in addition to Standard of Care (steroid therapy with or without additional therapies) .

At the conclusion of the dose escalation segment of the study, if the 300 mg Cannabidiol dose level/placebo is deemed safe for two weeks with Standard of care dose of steroids, patients will continue receiving this 300 mg dose/placebo for an additional period of 3 months. Weekly tapering off of steroids will then commence and will be carried out .

Three months after starting treatment with Cannabidiol an interim analysis to evaluate Cannabidiol's safety and efficacy will be carried out and treatment assignment group may be changed (according to response confirmation)

DETAILED DESCRIPTION:
Individual patient Standard of Care (steroid therapy with or without additional therapies) will be administered in a stable fashion during the first weeks of the study in addition to increasing doses of Cannabidiol or placebo ( in a double blind manner. Dosage of Cannabidiol will start at 25 mg twice a day and will be increased every two days, if no side effects are observed, to 50 mg twice a day, 100 mg twice a day and finally to 150 mg twice a day Cannabidiol respectively. Treatment will be given with food. Identical placebo will be administered in the placebo arm. In stage 1,both patient and investigator will be blinded to treatment modalities.

At the conclusion of the dose escalation segment of the study, if the 300 mg Cannabidiol dose level/placebo is deemed safe for two weeks with Standard of care dose of steroids, patients will continue receiving this 300 mg dose/placebo for an additional period of 3 months. Weekly tapering off of steroids will then commence and will be carried out .

Three months after starting treatment with Cannabidiol an interim analysis to evaluate Cannabidiol's safety and efficacy will be carried out by an independent assessor not associated with the study .At the conclusion of this interim analysis, Cannabidiol Non-responders will be removed from the trial, and Placebo Non-responders will be switched over to Cannabidiol.

If a patient flares, then his/her code will be opened by the unblinded observer. If the subject has been administered placebo, then he/she will be crossed over to the Cannabidiol arm. If the subject has been administered Cannabidiol, then he/she will be restarted on Standard of care prednisone in addition to Cannabidiol or removed from study, depending on the severity of the flare-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy confirmed, active, steroid dependent CD, without nutrient absorbance problems (Definition of steroid dependency: CD being treated with at least 5 mg/day steroids for the last 3 months; an attempt to reduce the dose induces flare of disease as determined by physician assessment).
2. Age ≥18 years
3. Steroid treatment of at least 3 months and stable steroid dose for at least 2 weeks .If thiopurines and/or biologics are also being administered, then must be administered at stable dose(s) for at least 3 months.
4. Patients will undergo an ECG and QT parameters will be measured for further analysis.
5. Female subjects who are postmenopausal (absence of menses for ≥ 2 years confirmed by a follicle stimulating hormone test), or who are surgically sterilized may be enrolled. Similarly, women of childbearing potential who had a negative pregnancy test at screening, who are willing to use two medically acceptable methods of contraception for the duration of the study as well as for at least three months after cessation of CBD treatment and who are willing to undergo pregnancy testing according to the study protocol may be enrolled.
6. Female subjects who are not breast-feeding and who have no intention to breast-feed during the term of the trial and for at least three months after cessation of CBD treatment may be enrolled.
7. Subject able to provide written informed consent

Exclusion Criteria:

1. Viral Hepatitis (HAV, HBV, HCV)
2. HIV
3. Serious psychiatric or psychological disorders
4. Active consumption of illicit drugs including cannabis or derivatives for at least 3 months prior to the study
5. Patients with short bowel syndrome, symptomatic stricture, abscess, recent history (within the previous 3 months) of abdominal surgery, nutrient absorbance problems
6. Patients whose disease is inaccessible by endoscopy
7. Patients with significant cardiac, respiratory or active malignance disease (except Basel Cell Carcinoma) comorbidities.
8. Any uncontrolled infection at time of registration
9. Renal comorbidity: eGFR < 30 mL/min/1.73 m2 (note: CKD Grade 4 is defined as eGFR 15-29 mL/min/1.73 m2)
10. Patient who is taking immunomodulatory medications for other indication
11. Women of child-bearing potential who intend to become pregnant or who are pregnant or breastfeeding

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of up to 300 mg CBD/day measured by Adverse Events | 12 month
  significance of the difference in percent of subjects experienced any Adverse events, drug-related Adverse events and Serious Adverse events between the study groups
Efficacy will be mesursed by precentegae of reduction in dose of steroids without flares | 12 month
  50% reduction in dose of steroids without flares

SECONDARY OUTCOMES:
Percentage of patients without flares | 12 month
  Disease flare will be recorded during the study
Percent of patients who did not demonstrate an increase in inflammatory activity | 12 month
  inflammatory activity scored will be measured during the study

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba
  - Shamir Medical Center, Tzrifin

IPD SHARING:
Plan to Share IPD: No